CLINICAL TRIAL: NCT00658827
Title: Exposure to Remicade (Infliximab) During Pregnancy in Patients With Inflammatory Bowel Disease, Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis and Psoriasis: a Review and Analysis of Birth Outcomes From the Swedish, Danish and Finnish Medical Birth Registers
Brief Title: Analysis of Birth Outcomes of Swedish, Danish and Finnish Women Exposed to Remicade With Inflammatory Bowel Disease, Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Psoriasis
Status: Completed | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013141; C0168T71 (Other: Janssen Biotech, Inc.)
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Psoriasis; Pregnant women exposed to infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group 1a: Remicade Cohort: Female patients who were exposed to Remicade at any time during pregnancy (and up to 3 months prior to LMP, if this information is available).
  Interventions: Other: No intervention
- Group 1b: Remicade Cohort: Infants born to Group 1a patients.
  Interventions: Other: No intervention
- Group 2a: Other Anti-TNF agents Cohort: Female patients who were exposed to anti-TNFs other than Remicade at any time during pregnancy (and up to 3 months prior to LMP, if this information is available).
  Interventions: Other: No intervention
- Group 2b: Other Anti-TNF agents Cohort: Infants born to Group 2a patients.
  Interventions: Other: No intervention
- Group 3a: Non-biologic Systemic Therapy Control Cohort: Female patients who were exposed to systemic therapy other than biologic agents at any time during pregnancy (and up to 3 months prior to LMP, if this information is available).
  Interventions: Other: No intervention
- Group 3b: Non-biologic Systemic Therapy Control Cohort: Infants born to Group 3a patients.
  Interventions: Other: No intervention
- Group 4a: Population Control Cohort: Female patients with no record of the diseases of interest and no exposure to biologic or non-biologic systemic therapy at any time during pregnancy (and up to 3 months prior to LMP, if the information is available).
  Interventions: Other: No intervention
- Group 4b: Population Control Cohort: Infants born to Group 4a patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. Patients receiving infliximab or anti-TNF as per the prescribing information will be observed.

SUMMARY:
The purpose of this study is collection and analysis of information pertaining to pregnancy outcomes in women exposed to infliximab during pregnancy, relative to the background risk in similar but non-biologic exposed patients; and information pertaining to health status, during the first year following delivery, of infants born to women following prenatal exposure to infliximab and their unexposed counterparts.

DETAILED DESCRIPTION:
This registry will analyze birth outcomes data from Medical Birth Registers on approximately 370 women who have become pregnant and have been exposed to infliximab with the diseases of interest: Inflammatory Bowel Disease (Crohn's Disease [CD] and Ulcerative Colitis [UC]), Rheumatoid Arthritis [RA], Psoriatic Arthritis [PsA], Ankylosing Spondylitis [AS], and Psoriasis (Pso) as well as all women with the same diseases who have not been exposed to infliximab. Demographics and information related to the diseases of interest, past medical history, infliximab exposure during pregnancy (and up to 3 months prior to conception), use of other medications, and pregnancy outcomes information and infant birth information will be collected from the Swedish national health registries (a. Swedish Medical Birth Register [SMBR] b. Swedish Prescribed Drug Register c. Swedish Patient Register [PAR]), Danish national health registries (a. Danish Medical Birth Register [DMBR] b. Danish Register of Medicinal Product Statistics c. Danish National Patient Registry), and Finnish national health registries (a. Finnish Medical Birth Register [FMBR] b. Finnish Register on Prescribed Medicine c. Finnish National Care Register for Health Care Institutions [HILMO] d. Finnish Register on Congenital Malformations) during the study period. The health status of infants born to these women will be followed for 1 year after birth. During the 1-year follow-up period, information related to hospitalizations and antibiotic use will be obtained. No study medications will be administered in this registry. Treatments are as prescribed by the physician on the basis of usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Study patients must meet the following criteria: Women of childbearing age with birth outcomes recorded in either the Swedish Medical Birth Register (SMBR), Finnish Medical Birth Register (FMBR) or in the Danish Medical Birth Register (DMBR) who have confirmed diagnosis of Crohn's disease, ulcerative colitis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or psoriasis and documented exposure to infliximab during pregnancy and infants born to these women
* Control patients must meet the following criteria: Women of childbearing age with birth outcomes recorded in either the SMBR, FMBR or DMBR who have confirmed diagnosis of Crohn's disease, ulcerative colitis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis or psoriasis, and no exposure to biologics during pregnancy and infants born to these women

Exclusion Criteria:

* Information for women who do not have a documented history of the diseases of interest but whose birth outcomes are included in the SMBR, FMBR or DMBR during the study period and the infants of these women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Female patients of child bearing age with one of the diseases of interest and infants delivered by such patients.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Number of normal live birth observed in pregnant women exposed and not exposed to infliximab | 5 years
Number of abnormal live birth observed in pregnant women exposed and not exposed to infliximab | 5 years
  Abnormal live birth will be considered if the birth outcome is preterm birth, small for gestational age/intrauterine growth retardation, malformations, or perinatal morbidity.
Number of fetal death observed in pregnant women exposed and not exposed to infliximab | 5 years
Number of normal live birth observed in pregnant women with disease entity of interest exposed and not exposed to infliximab | 5 years
Number of abnormal live birth observed in pregnant women with disease entity of interest exposed and not exposed to infliximab | 5 years
  Abnormal live birth will be considered if the birth outcome is preterm birth, small for gestational age/intrauterine growth retardation, malformations, or perinatal morbidity.
Number of fetal death observed in pregnant women with disease entity of interest exposed and not exposed to infliximab | 5 years

SECONDARY OUTCOMES:
Antibiotic use and hospital care during the first year after birth for infliximab exposed and non-exposed infants | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.